CLINICAL TRIAL: NCT06673758
Title: Effects of Taichi Exercises on Cardiorespiratory Fitness Among School Going Childern
Brief Title: Effects of Taichi Exercises on Cardiorespiratory Fittness
Acronym: taichi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0712
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Child, Only
Keywords: cardiorespiratory fitness,exercise ,pediatrics,tai chi.
MeSH Terms: interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Intervention Model Description: parallel assignment It will be randomized control trail in which non probality convienent sampling will b used.two groups of 10 to 14 years will be formed in which participants randomly diveded.group one receive art and crafts activity and other receive tai chi exercises of two weeks sessions
Who Masked: Participant
Masking Description: participants will get seperate treatment protocols and possible efforts will be put to mask the both group about treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): experimental group given tai chi exercises on three levels of two weeks sessions of total 10 session in five days of each week.
  Interventions: Other: tai chi exercises
- control group (Other): 15 participants are given art and crafts activity of two weeks
  Interventions: Other: Art and crafts activity

INTERVENTIONS:
Other: tai chi exercises — tai chi exercises of three basic levels will be given with sessions of two weeks five time a day and follow efftects of tai chi exercises by 6minute walk test and time up and go test and check the results before and after exercises
  Other Names: art and crafts activity
  Arms: experimental group
Other: Art and crafts activity — Art and crafts activity will be given to control group and check cardiorespiratory fitness before and after arts and crafts activity
  Arms: control group

SUMMARY:
Effects of tai chi exercises on cardiorespiratory fitness among scchool going childern. sample size is 30 .divided two groups into 15 15 members one group is giving hand and art crafts activity other is giving tai chi basics level exercises then check and compare cardiorespiratory fitness by time up and go test and 6 minutes walk test. compare the results.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial involving 30 participants, with data collected from the Sanai school system in Sargodha. The study will include school-aged children with normal weight between the ages of 10 and 14. Children with any cardiorespiratory conditions, hemophilia, muscular dystrophy, or a history of cardiovascular events will be excluded. The sample of 30 will be divided into two groups of 15 participants each. Group A will participate in tai chi exercises across three levels, while Group B will engage only in basic arts and crafts activities. The interventions will consist of 10 sessions, conducted at a rate of 5 sessions per week over 2 weeks. To assess the respiratory fitness of the children, data will be collected using the 6-minute walk test and the Timed Up and Go test. Data analysis will be performed using SPSS version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* childerns with 10 to 14 years
* childerns with normal weight less than 30kg/m2

Exclusion Criteria:

* Childerns with any cardiorespiratory issues
* Childerns who have gone through CVA,hemophilia, dystrophy and conditions which impact cardiorespiratory status

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | 2 weeks
  6 minutes walk test is use for diagnosis of cardiorespiratory fitness after tai chi and art andcrafts activity

SECONDARY OUTCOMES:
time up and go test | 2 weeks
  time up and go test will be use after tai chi exercises and art and crafts activity

CONTACTS AND LOCATIONS:
Overall Officials: Anum Saleem, MS*, Principal Investigator — Ripah International university
Locations (2):
- Pakistan (2):
  - Riphah international university, Lahore, Punjab Province
  - Imran Amjad, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Tian J, Yang Q. Tai Chi exercise improves working memory capacity and emotion regulation ability. Front Psychol. 2023 Feb 17;14:1047544. doi: 10.3389/fpsyg.2023.1047544. eCollection 2023. PMID 36874821